CLINICAL TRIAL: NCT06845176
Title: Comparison of Three Modalities of Combining Motor Imagery and Tendon Vibration on the Effectiveness of Motor Imagery
Brief Title: Combining Motor Imagery and Tendon Vibration on the Effectiveness of Motor Imagery
Acronym: IMVT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Jean Monnet University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24CH250; 2024-A02856-41 (Other: ANSM)
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteer
Keywords: Kinesthetic motor imagery; Tendon vibration; Corticospinal excitability; Neuroplasticity; Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Simultaneous application of TV and kMI (Experimental): Simultaneous application of Tendon Vibration and Kinesthesic Motor Imagery
  Interventions: Device: Tendon vibration (TV); Other: Kinesthetic motor imagery (kMI)
- TV application between kMI trials (Experimental): Tendon Vibration application between Kinesthesic Motor Imagery
  Interventions: Device: Tendon vibration (TV); Other: Kinesthetic motor imagery (kMI)
- TV as a pre-conditionning for kMI (Experimental): Tendon Vibration application as a pre-conditionning for Kinesthesic Motor Imagery
  Interventions: Device: Tendon vibration (TV); Other: Kinesthetic motor imagery (kMI)

INTERVENTIONS:
Device: Tendon vibration (TV) — We use the VIBRAMOOV PHYSIO device which delivers local muscle vibrations at frequencies of 80 Hz and an amplitude of 1 mm.
Other: Kinesthetic motor imagery (kMI) — kMI is a mental technique in which an individual visualizes performing a movement without physically executing it. This process involves the internal representation of the sensations associated with the movement, engaging neural pathways similar to those activated during actual physical movement. kMI stimulates key motor and sensory areas in the brain, promoting neuroplasticity and enhancing motor performance.

SUMMARY:
Kinesthetic motor imagery (kMI) involves imagining the sensations of movement, activating brain regions similar to actual movement execution. It is widely used to maintain or restore motor functions, particularly in rehabilitation. Tendon vibration (TV), which stimulates proprioceptive receptors can also enhance corticospinal excitability and promote neuroplasticity. This project investigates the coupling of kMI and TV through three modalities: simultaneous application, TV application between kMI trials, or pre-application of TV to precondition the nervous system before kMI trials. The effectiveness and quality of kMI will be assessed by corticospinal excitability measurements using transcranial magnetic stimulation and EEG measures. Conducting this study in healthy participants will inform the development of optimized clinical interventions for immobilized or mobility-reduced patients.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 50 years.
* Affiliated with or beneficiaries of a social security system.
* Provided written informed consent freely after being informed of the study's purpose, procedures, and potential risks.

Exclusion Criteria:

* History of pathology or surgery affecting upper limb motor function within 6 months prior to the study.
* Chronic neurological, motor, or psychiatric disorders.
* Use of neuroactive substances likely to alter corticospinal excitability (e.g., hypnotics, antiepileptics, psychotropics, muscle relaxants) during the study period.
* Contraindications to transcranial magnetic stimulation
* Simultaneous participation in another interventional study or participation in such a study within 30 days prior to this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-03-11 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Optimization of kMI | 30 minutes
  We will measure corticospinal excitability. This will be assessed by the area (in mV.%) under the curve representing the amplitude of motor-evoked potentials (MEPs, in mV) recorded via electromyography, as a function of transcranial magnetic stimulation intensity (in % of the stimulator's maximal output) required to evoke these potentials.

CONTACTS AND LOCATIONS:
Overall Officials: Léonard FEASSON, PhD, Principal Investigator — Centre Hospitalier Universiatire de SAINT-ETIENNE
Locations (1):
- IRMIS-Hôpital Nord, Saint-Etienne, France, France

IPD SHARING:
Plan to Share IPD: No
This study is being conducted in a single department of the ST-ETIENNE University Hospital.